CLINICAL TRIAL: NCT02208128
Title: Molecular Determinants for Therapy Response on Renal Cell Carcinoma
Acronym: MORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-539/2013; DRKS00006193 (Other: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2014-06-02; First posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Biomarkers; Molecular modifications
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; pazopanib; Bevacizumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Receptor-Tyrosinkinase-Inhibitor (No Intervention): Guidelines-oriented therapy with approved systemic medications for renal cell carcinoma individually for each patient (Receptor-Tyrosinkinase-Inhibitor) (e.g.Sunitinib, Pazopanib, Bevacizumab, Everolimus, Axitinib, Temsirolimus). With 1.progression turning to second line treatment with one of the upper mentioned medications. Third line therapy due to the individual molecular modifications for each patient.
  Interventions: Drug: Sunitinib, Pazopanib, Bevacizumab, Everolimus...

INTERVENTIONS:
Drug: Sunitinib, Pazopanib, Bevacizumab, Everolimus... — Clinical standard
  Other Names: e.g.Sunitinib, Pazopanib, Bevacizumab, Everolimus...

SUMMARY:
Aim of the scientific analysis is to find biological factors (biomarkers) allowing a prediction of disease progression and a better choice of therapy. After diagnosis the kidney and the tumor will be removed by standard surgery followed by drug therapy. Within surgery remaining tumor tissue will be used for the scientific analysis. In case of disease progression during the drug treatment the drug therapy will be changed. Before therapy change a small tissue sample will be collected for molecular diagnostics. This will be done by puncture through the skin under local anesthesia. Blood samples taken before surgery and at the time of first and second disease progression will also be used for molecular-biological analysis. As there is no clear recommendation for drug therapy after disease progression this study should serve to determine an individual therapy on the basis of the molecular profile and the molecular changes. As the tumor disease changes and developes resistance to drugs, analysis at the time of disease progression shall identify biological factors which will predict a likelihood response to a specific drugs.

This shall allow to give the patient an individual therapy.

DETAILED DESCRIPTION:
Aim of this study is to perform a profound molecular analysis of the tumor before beginning therapy and after failure of the approved targeted first-and second line therapy (standard therapy). The tumor sample will be analyzed by using profound molecular analysis to identify target structures which will predict the efficacy of a specific therapy (substance group)and therefore have a predictive value. The analysis of molecular biomarkers include the genomic sequencing of targeted areas or of the entire DNA of the tumor tissue comparative to the DNA of healthy cells, the measurement of DNA-regulatory elements (methylation, mi-RNA expression, protein expression analytics, functional tumorcell analysis in-vitro, efficacy analysis in cell culture or in animal model) who are supposed to inspect the biological influence of the molecular biomarkers and measurements of free tumor DNA out of the blood.

The response to the established standard therapy in the first and second line will be acquired due to all clinical and radiological established standard parameters. The clinical-radiological response will be correlated with the molecular changes and their changes in therapy process to allow predictive prognosis for a further therapy.

There is no approved clinical standard for third line therapy. However there are further medications approved without any scientific evidence of their efficacy in this therapy situation (third line treatment after failure of first and second line treatment) and for which a response of under 6 weeks is expected.

For these patients the third line therapy will be adjusted to the molecular profiles of the previous therapies. Therefore the oncological history of the noticed marker profiles and the presence of target structures (from whom it is known that they are influenced by certain substances) will be considered.

The therapy will use substances which are approved in general for the treatment of metastatic renal cell cancer.

ELIGIBILITY:
Inclusion Criteria:

Minimum Age: 18 Years Maximum Age: no maximum age

* metastatic lesions easy of access for puncture for specimen storage
* histological subtype: clear-cell renal cancer
* no contraindications against systemic therapy
* indication for systemic therapy given

Exclusion Criteria:

* preexisting mental illness
* further active malignancy
* patients with increased risk of bleeding and/or wound healing disorder
* patients who are not legally competent or unable to consent
* contraindication for surgical intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression in third line therapy | Approximately 2 years depending on when the failure in third line therapy happens
  Progression free survival in third-line therapy ( defined as the time from beginning of the third-line therapy to the date of the first documented progression as determined by the investigator using Response Evaluation Criteria in Solid Tumors criteria assessed by CT/MRI every 12 weeks).

SECONDARY OUTCOMES:
Identification of preventive biomarkers. | 2weeks in average before surgery and 4 weeks in average after surgery before starting first line treatment
  Identification of preventive biomarkers.

OTHER OUTCOMES:
Identification of preventive biomarkers | 2years

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Pahernil, PD Dr., Principal Investigator — University of Heidelberg, Urological Department
Locations (1):
- Urological Department of the University Hospital Heidelberg, Heidelberg, Germany